CLINICAL TRIAL: NCT02141789
Title: Outpatient Psychotherapeutic Treatment for Alcohol Dependent Individuals With Comorbid Psychiatric Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Konstanz (Other)
Responsible Party: Principal Investigator, Michael Odenwald, Dr. rer. nat., Dipl. Psych., Licensed Psychotherapist, University of Konstanz
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UKonstanzMOdenwald2014-1
Record Dates: First submitted 2014-05-15; First posted 2014-05-19 (Estimated); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Alcohol Dependence
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Outpatient Cognitive Behavioral Psychotherapy (Experimental): Outpatient Cognitive Behavioral Therapy is a well-known and frequently applied psychotherapy approach that does not need further description.
  Interventions: Behavioral: Outpatient Cognitive Behavioral Psychotherapy

INTERVENTIONS:
Behavioral: Outpatient Cognitive Behavioral Psychotherapy — Integrated CBT intervention for alcohol dependence and comorbid psychiatric disorder (we include only patients with comorbid mood or anxiety disorders).
Behavioral: Outpatient Cognitive Behavioral Psychotherapy — The intervention is a well established form of psychotherapy that has infrequently been used in the German system with this group of patients in contrast to many other countries where it is the standard approach, e.g. the US.

SUMMARY:
Research has shown that alcohol dependence often co-occurs with comorbid anxiety disorders and/or depression. Anxiety and depression influence the course and treatment of alcohol dependence and are a major risk factor for alcohol relapse within the first three months after detoxification. Therefore, there is need for combined treatment (integrated therapy) of alcohol dependence and comorbid psychiatric disorders, e.g. anxiety and/or depression. Until today, there are no systematic outpatient treatment offers for this special group of patients in Germany. In this study we want to investigate if integrated outpatient cognitive behavioral therapy can prevent and decrease alcohol relapse within the first three months after detoxification. Therefore we hypothesize that immediate start of integrated outpatient psychotherapy will reduce relapse variables compared to treatment as usual which is characterized by non-immediate start of therapy due to the required application for insurance coverage.

ELIGIBILITY:
Inclusion Criteria:

* alcohol dependence
* comorbid anxiety or mood disorder

Exclusion Criteria:

* severe mental illness: psychosis, mania, personality disorders
* current suicidality
* non-compliance with appointments during first 5 sessions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Relapse | 3 months
  We assess whether participants have an alcohol relapse (any drinking of alcohol) in the three months after study inclusion
Days with heavy alcohol drinking | 3 months
  We assess with the Timeline Follow Back (TLFB, Sobell & Sobell, 2000) the number of days with heavy alcohol drinking (for a man 5 or more drinks a day, for a woman 4 or more drinks a day) in the three months after study inclusion

SECONDARY OUTCOMES:
Comorbid psychiatric symptoms | 3 months
  Anxiety, depression and other relevant psychiatric symptoms will be measured by different standardized questionnaires at t1 (before treatment) and after 3 months (t2). We will use standardized symptom change as outcome measure.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Odenwald, Dr. rer. nat., Principal Investigator — University of Konstanz
Locations (1):
- University of Konstanz, Outpatient Clinic for Psychotherapy, Konstanz, Germany

REFERENCES:
- [Result] Schawohl A, Adam M, Odenwald M. What's Next After Withdrawal Treatment? A Randomized Controlled Pilot Study on Integrated Outpatient Psychotherapy in Alcohol-Dependent Patients With Dual Diagnoses. Zeitschrift für Klinische Psychologie und Psychotherapie. 2018; 47(3): 153-162. doi: 10.1026/1616-3443/a000487